CLINICAL TRIAL: NCT04156386
Title: The Effect of Vegan or Animal Protein Ingestion on the Recovery of Skeletal Muscle Function Following Strenuous Exercise
Brief Title: Vegan or Animal Protein Ingestion on the Recovery of Muscle Function Following Exercise
Acronym: VAMPIRE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Exeter (Other)
Collaborators: Beachbody (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Other
Other Study IDs: 190703-B-01
Record Dates: First submitted 2019-09-06; First posted 2019-11-07 (Actual); Last update posted 2023-03-22 (Actual); Status verified 2023-03

CONDITIONS: Muscle Recovery
Keywords: Muscle Strength; Musculoskeletal Physiology; Muscle, Skeletal; Whey Proteins; Plant Proteins; Dietary supplements
MeSH Terms: interventions — Whey; maltodextrin

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Animal Protein (Active Comparator)
  Interventions: Dietary Supplement: Recovery animal (20g whey) protein supplement
- Vegan Protein (Active Comparator)
  Interventions: Dietary Supplement: Recover vegan (26g pea) protein supplement
- Placebo (Placebo Comparator)
  Interventions: Dietary Supplement: Placebo (32g maltodextrin)

INTERVENTIONS:
Dietary Supplement: Recovery animal (20g whey) protein supplement — Animal protein supplement consumed post exercise to aid recovery of muscle function following strenuous exercise.
  Arms: Animal Protein
Dietary Supplement: Recover vegan (26g pea) protein supplement — Vegan protein supplement consumed post exercise to aid recovery of muscle function following strenuous exercise.
  Arms: Vegan Protein
Dietary Supplement: Placebo (32g maltodextrin) — Placebo consumed post exercise to aid recovery of muscle function following strenuous exercise.
  Arms: Placebo

SUMMARY:
This study will assess the effect of daily post-exercise vegan (pea) and animal (whey) protein ingestion compared to placebo over 7 days of recovery from strenuous exercise. Muscle strength and soreness will be measured daily, and mechanisms underpinning recovery will be investigated in muscle biopsies taken 3, 24 and 48 hours after exercise.

DETAILED DESCRIPTION:
Strenuous exercise can cause muscle soreness and reduced muscle strength. It is widely acknowledged that nutritional supplements derived from animal protein sources, including whey from milk, aids recovery when taken immediately after strenuous exercise. However, the effect of vegan protein supplements are less understood, and how they affect recovery of strength and soreness is not known. This is an important area of research due to the increasing demand for plant-based protein.

ELIGIBILITY:
Inclusion Criteria:

* Recreationally active
* 18-40 years of age

Exclusion Criteria:

* Regular and structured involvement in resistance training
* Inactive participants
* Habitual dietary protein intake <0.8g/kg bw/day and >2.0g/kg bw/day
* Use of nutritional supplements
* Any diagnosed metabolic conditions (diabetes), cardiovascular disease or hypertension
* Current musculoskeletal injury
* Use of anti-inflammatory medicines
* Individuals with non -removable metallic implants (including heart pacemaker, cochlea implants, medication pumps, surgical clips, plates or screws) or claustrophobia
* Individuals with an allergy to egg, fish, wheat or soy ingredients as the product is manufactured in a facility that contains these ingredients

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 30 (Actual)
Dates: Start 2019-09-23 (Actual); Primary Completion 2022-04-23 (Actual); Study Completion 2022-04-23 (Actual)

PRIMARY OUTCOMES:
Change in isokinetic work (W30) performed before and every 24 h after performing 300 maximal eccentric quadriceps contractions. | Once per 24 hour period for 7 days
  The recovery of skeletal muscle isokinetic force production following eccentric exercise using an isokinetic dynamometer

SECONDARY OUTCOMES:
Perceived quadriceps muscle soreness | Once per 24 hour period for 7 days
  Soreness will be assessed using a visual analogue scale (VAS) to determine whether the protein supplement can reduce muscle soreness following eccentric exercise. This scale will represent a 100mm line with no pain and worst pain anchored at either end of the scale.
Muscle swelling | Once per 24 hour period for 3 days
  Determine whether the protein supplement can reduce muscle swelling following eccentric exercise assessed using MRI
Rate of protein incorporation into the muscle | Once per 24 hour period for 3 days
  Determine whether the strenuous exercise and a protein supplement can upregulate protein synthesis following strenuous exercise assessed by muscle biopsies
Plasma creatine kinase (CK) activity before and every 24 h after performing 300 maximal eccentric quadriceps contractions. | Once per 24 hour period for 7 days
  Damage and inflammatory bio markers following strenuous exercise assessed by blood sample
Change in flow mediated dilation | Once hourly post exercise for 3 hours
  Determine whether the protein polyphenol supplement can impact vascular function following eccentric exercise

CONTACTS AND LOCATIONS:
Overall Officials: Francis Stephens, Principal Investigator — University of Exeter
Locations (1):
- University of Exeter, Exeter, United Kingdom

IPD SHARING:
Plan to Share IPD: No